CLINICAL TRIAL: NCT00200564
Title: Ketamine and Postoperative Analgesia in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: BRD/03/12-H
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2005-07

CONDITIONS: Postoperative Analgesia
Keywords: Pediatrics; ketamine; postoperative analgesia; nalbuphine; Postoperative analgesia in children
MeSH Terms: interventions — Ketamine

INTERVENTIONS:
Drug: ketamine

SUMMARY:
The benefit of small doses of ketamine has been demonstrated for postoperative analgesia in adults but remains unproved in children. The investigators' purpose is to evaluate the effects of continuous intravenous small doses of ketamine versus placebo to improve the quality of postoperative analgesia in children (6 months to 6 years of age). Caudal anesthesia is performed for intraoperative analgesia and all children receive paracetamol, a non-steroidal anti-inflammatory and continuous intravenous nalbuphine.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 months to 6 years of age
* American Society of Anesthesiologists (ASA) I or II
* Undergoing elective surgery with intraoperative caudal analgesia

Exclusion Criteria:

* ASA III or IV
* Contraindication to caudal anesthesia
* Allergy to drugs used in the study
* Failure in caudal puncture
* Administration of morphine derivative

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2004-02

PRIMARY OUTCOMES:
Area under the curve of pain scores (CHEOPS) measured | every 2 hours during the first 24 hours after eyes open

SECONDARY OUTCOMES:
Evaluation by the parents and nurses of the quality of analgesia with a visual analogue scale graded from 0 to 10 | at the 24th hour
Number of painful episodes requiring additional boluses of nalbuphine
Number of children requiring morphine after inefficiency of additional boluses of nalbuphine
Percentage of children with side effects related to injection of ketamine
Time to complete feeding
Percentage of children with nausea or vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Bazin, MD, Principal Investigator — Nantes UH
Locations (1):
- Nantes University Hospital, Nantes, France